CLINICAL TRIAL: NCT00109772
Title: A Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lenalidomide in the Treatment of Complex Regional Pain Syndrome Type 1
Brief Title: Study to Evaluate the Efficacy and Safety of Lenalidomide in the Treatment of Complex Regional Pain Syndrome Type 1
Acronym: CRPS-002
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis showed the primary outcome was not reached
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-CRPS-002
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Complex Regional Pain Syndrome, Type I
Keywords: CRPS; RSDS; Pain; CC-5013; Revlimid; Complex Regional Pain Syndrome; Reflex Sympathy Dystrophy Syndrome; Lenalidomide; CRPS Type I; Celgene
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Pain; Complex Regional Pain Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lenalidomide (Experimental): 10 mg/day lenalidomide orally for up to 12 weeks in the double-blind treatment period. Participants who completed double-blind treatment had the option of continuing on lenalidomide in the open-label extension period for as long as benefit was derived from the drug or until study closure.
  Interventions: Drug: lenalidomide
- Placebo (Placebo Comparator): Placebo orally for up to 12 weeks in the double-blind treatment period. Participants who completed double-blind treatment had the option of crossing over to lenalidomide 10mg in the open-label extension period for as long as benefit was derived from the drug or until study closure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lenalidomide — Two 5 mg capsules taken one time per day
  Other Names: Revlimid; CC-5013
  Arms: lenalidomide
Drug: Placebo — Two placebo capsules taken one time per day
  Arms: Placebo

SUMMARY:
The purpose of this multicenter, double-blind, placebo-controlled study is to evaluate the efficacy and safety of Lenalidomide in adult subjects with Complex Regional Pain Syndrome (CRPS) Type 1.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled study in adult subjects with Complex Regional Pain Syndrome (CRPS) Type 1.

One hundred eighty (180) subjects diagnosed with unilateral CRPS Type 1 will be enrolled and randomized to receive orally either 10 mg/day of lenalidomide or placebo (90 subjects per treatment arm). For each subject, the study consists of three phases: Pre-randomization Phase (2 weeks), Treatment Phase (12 weeks) and Extension Phase where subjects have the opportunity to receive lenalidomide treatment as long as a benefit is derived from the drug. Subjects who complete all 12 weeks of the treatment phase may be eligible to receive lenalidomide in the extension phase. Subject may continue in the extension phase as long as a benefit is derived from the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at the time of signing the informed consent form
* Understand and voluntarily sign an informed consent form
* A diagnosis of CRPS Type 1, as defined by modified International Association for the Study of Pain criteria for at least a one-year duration. Unilateral involvement of a distal limb (hand or foot) with or without proximal spread must be present. In the presence of upper and lower limb involvement, the most severely affected limb will be designated the CRPS-affected limb.
* Screening: CRPS pain intensity score in the CRPS-affected limb must be at least 4 on an 11-point (0-10) Pain Intensity Numerical Rating Scale (PI-NRS).
* Randomization: Average PI-NRS score for randomization purposes will be based on AM and PM assessments made during the 7 days prior to randomization. At least eight PI-NRS scores during this 7-day period are required and the Average PI-NRS score in the CRPS-affected limb during this period must be at least 4 on an 11-point (0-10) PI-NRS.
* Measurable (by electrophysiology methods) sural, median sensory, median motor and peroneal motor nerves at the screening nerve conduction study.
* Opioid analgesics, non-opioid analgesics, non-steroidal anti-inflammatory drugs, anticonvulsants, antidepressant drugs and other non-drug therapies may be continued provided that the subject is on stable doses/regimens for at least four weeks prior to the start of the Treatment Phase (Visit 2).
* Able to adhere to the study visit schedule and other protocol requirements.
* Women of childbearing potential (WCBP) must agree to practice complete abstinence from heterosexual intercourse or to use two methods of contraception beginning 4 weeks prior to the start of study drug (Day 1) while on study drug (including dose interruptions) and 4 weeks after the last dose of study drug. The two methods of contraception must include one highly effective method (i.e. intrauterine device [IUD], hormonal [birth control pills, injections, or implants only if used in conjunction with a low-dose (81 mg/day) aspirin regimen], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). If a hormonal method (birth control pills, injections, or implants) or IUD is not medically possible for the subject, two of the barrier methods will be acceptable.
* Women of childbearing potential (WCBP) must have two negative pregnancy tests (sensitivity of at least 50 mlU/mL) prior to starting study drug treatment. The first test should be performed within 10-14 days and the second within 24 hours of starting study drug. Once treatment has started, it is recommended that subjects have weekly pregnancy test during the first 4 weeks of treatment. Thereafter, subjects are required to have pregnancy testing every 4 weeks in females with regular menstrual cycles and every 2 weeks in females with irregular cycles.
* Males (including those who have had a vasectomy) must use barrier contraception (latex condoms) when engaging in reproductive sexual activity with WCBP while on study drug and for 4 weeks after the last dose of study drug.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

* History of deep vein thrombosis (DVT) or stroke in the past 5 years.
* Documented peripheral neuropathies to include diabetic neuropathy and other metabolic or toxic neuropathies.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Any other serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* White blood cell count (WBC) < 3.5*10^9/L at screening.
* Bilirubin, alanine transaminase (ALT), aspartate transaminase (AST) or alkaline phosphatase levels more than two times the upper limit of the normal range at screening.
* Abnormal thyroid function test values at screening.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of concomitant medication(s), which could increase the risk for developing DVT, except for steroid-based contraceptives (oral injectable, implantable) and hormone replacement therapies only if used in conjunction with a low-dose (81 mg/day) aspirin regimen.
* Concurrent use of thalidomide.
* Prior development of an allergic reaction/hypersensitivity while taking thalidomide.
* Prior development of a moderate or severe rash or any desquamation while taking thalidomide.
* Prior treatment with lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2005-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Manning, MD, PhD, Study Director — Celgene Corporation
Locations (27):
- United States (27):
  - Pivotal Research Centers, Peoria, Arizona
  - UCSD Center for Pain and Palliative Medicine, La Jolla, California
  - Loma Linda Institution, Loma Linda, California
  - Space Coast Neurology, Palm Bay, Florida
  - Northwestern University, Chicago, Illinois
  - Rehab Institute of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Pain Mgmt Ctr, St Louis, Missouri
  - Hospital for Joint Disease, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Hospitals University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Carolinas Pain Institute, P.A. & the Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Research Institute of Greater Dayton, Dayton, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Knobler Institute of Neurologic Disease, Fort Washington, Pennsylvania
  - Drexel University College of Medicine Department of Neurology Rm 7102, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech Medical Center Department of Anesthesiology, Lubbock, Texas
  - University of Virginia Pain Management Center, Charlottesville, Virginia
  - Swedish Pain Services, Seattle, Washington

REFERENCES:
- [Derived] Manning DC, Alexander G, Arezzo JC, Cooper A, Harden RN, Oaklander AL, Raja SN, Rauck R, Schwartzman R. Lenalidomide for complex regional pain syndrome type 1: lack of efficacy in a phase II randomized study. J Pain. 2014 Dec;15(12):1366-76. doi: 10.1016/j.jpain.2014.09.013. Epub 2014 Oct 2. PMID 25283471

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 184 participants were randomized to the study and 180 participants received at least 1 dose of study drug.
Groups:
- Placebo to Lenalidomide: Placebo orally for up to 12 weeks in the double-blind treatment period. Participants who completed double-blind treatment had the option of crossing over to lenalidomide 10mg in the open-label extension period for as long as benefit was derived from the drug or until study closure.
Period: Double-blind Treatment
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Started | 90 | 94
Safety and ITT Population | 87 (Safety: at least one dose of study drug ITT: treated and at least one post dose diary measurement) | 93 (Safety: at least one dose of study drug ITT: treated and at least one post dose diary measurement)
Completed | 68 | 79
Not Completed | 22 | 15
Not completed — Adverse Event | 14 | 5
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 0 | 4
Not completed — Withdrew prior to treatment | 3 | 1
Period: Open-label Extension
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Started | 64 (Four double-blind participants did not continue into the open-label extension) | 78 (One double-blind participant did not continue into the open-label extension)
Completed | 19 (Participants who were active in extension period when the sponsor terminated the study.) | 29 (Participants who were active in extension period when the sponsor terminated the study.)
Not Completed | 45 | 49
Not completed — Adverse Event | 10 | 19
Not completed — Lack of Efficacy | 19 | 11
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Other | 4 | 10

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Placebo to Lenalidomide | Total
Number analyzed (Participants) | 87 | 93 | 180
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (11.37) | 45.1 (11.06) | 44.5 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 79 | 144
  Male | 22 | 14 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  White | 81 | 86 | 167
  Black | 3 | 4 | 7
  Hispanic | 1 | 3 | 4
  Asian/Pacific Islander | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have a >= 30% Reduction (Improvement) in the Complex Regional Pain Syndrome (CRPS) Pain Intensity Numeric Rating Scale (PI-NRS) Score From Baseline to the Last Assessment
Description: Participants rated the intensity of pain in the CRPS-affected limb twice each day in a diary. The PI-NRS is an eleven point scale with 0=no pain and 10=worst pain imaginable. Responders are participants who completed 12 weeks of treatment and their week 12 PI-NRS score showed at least a 30% improvement from baseline. Participants who did not complete 12 weeks of treatment are considered non-responders.
Time Frame: Day 0, Week 12
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 87 | 93
percentage of participants
  Responders | 16.1 | 16.1
  Non-responders | 83.9 | 83.9
Statistical Analysis 1: Comparison: Lenalidomide vs Placebo to Lenalidomide; Test type: Superiority or Other; p = .8940, Cochran-Mantel-Haenszel; controlled for centers

2. Secondary Outcome: Change From Baseline in the Total Score of the Short Form McGill Pain Questionnaire (SF-MPQ) at Week 12
Description: Short Form McGill Pain Questionnaire (SF-MPQ) is comprised of 15 pain qualities that are rated by the participant on a 4 point scale with 0=none and 3=severe. The scale for the Total Score is 0-45. Week 12 values are compared to baseline values. Negative changes indicate improvement in level of pain.
Time Frame: Day 0, week 12
Population: Intent to treat. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | -5.2 (9.15) | -3.0 (9.37)

3. Secondary Outcome: Change From Baseline in the Complex Regional Pain Syndrome (CRPS) Pain Intensity Numeric Rating Scale (PI-NRS) Score Using Averaged Morning and Evening Readings at Week 12
Description: Participants rated the intensity of pain in the CRPS-affected limb twice each day in a diary. Morning and evening scores are averaged. The PI-NRS is an eleven point scale with 0=no pain and 10=worst pain imaginable. Week 12 values are compared to baseline values. Negative changes indicate improvement in level of pain.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | -0.6 (1.65) | -0.4 (1.50)

4. Secondary Outcome: Change From Baseline in the Morning Complex Regional Pain Syndrome (CRPS) Pain Intensity Numeric Rating Scale (PI-NRS) Score at Week 12
Description: Participants rated the intensity of pain in the CRPS-affected limb twice each day in a diary. The PI-NRS is an eleven point scale with 0=no pain and 10=worst pain imaginable. The morning pain ratings at baseline and Week 12 are compared. Negative changes indicate improvement in level of pain.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | -0.6 (1.67) | -0.4 (1.53)

5. Secondary Outcome: Change From Baseline in the Evening Complex Regional Pain Syndrome (CRPS) Pain Intensity Numeric Rating Scale (PI-NRS) Score at Week 12
Description: Participants rated the intensity of pain in the CRPS-affected limb twice each day in a diary. The PI-NRS is an eleven point scale with 0=no pain and 10=worst pain imaginable. The evening pain ratings at baseline and Week 12 are compared. Negative changes indicate improvement in level of pain.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | -0.6 (1.69) | -0.4 (1.53)

6. Secondary Outcome: Change From Baseline in Daily Sleep Assessment Average Score at Week 12
Description: Participants rated how much CRPS pain interfered with their sleep each day in a diary. The Sleep Assessment uses an eleven point scale for four questions. Questions concern ability to fall asleep, ability to stay asleep, how refreshed the participant feels upon waking and how alert the participant is during the day. All use a scale of 0-10, where the higher number is the positive response (e.g. 0=Pain completely interferes with sleep and 10=Pain does not interfere). The mean of all four responses was calculated if at least 3 of the 4 questions had a value. Week 12 values are compared to baseline values. Positive change values indicate improvement.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | 0.7 (1.48) | 0.7 (1.42)

7. Secondary Outcome: Change From Baseline in Activity Level Rating Using a Numeric Rating Scale (NRS) at Week 12
Description: Participants rated how the activity level on a given day compares with their activity level prior to the start of treatment. A seven-point scale is used with -3=much worse and +3=much better. Positive change values indicate improvement.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | 0.1 (1.08) | 0.2 (1.09)

8. Secondary Outcome: Change From Baseline in Participant Assessment of CRPS Symptoms Total Score at Week 12
Description: Participants rated twelve CRPS symptoms using a four-point rating scale in which 1=the most positive outcome and 4= the most negative outcome for a total scale of 12-48. Week 12 values are compared to baseline values. Negative change values indicate improvement.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Thirty-three participants had either no baseline or post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 67 | 80
units on a scale | -2.4 (6.27) | -1.4 (5.83)

9. Secondary Outcome: Change From Baseline in "Mechanically Evoked" (Allodynia) Numeric Rating Scale (NRS) Score at Week 12
Description: The investigator rated the degree of allodynia on both the CRPS-affected limb on an eleven-point scale where 0=no pain and 10=worst pain imaginable. This outcome compares the baseline values for the CRPS affected-limb to the values at week 12. Negative change values indicate improvement.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Sixteen participants had either no baseline or post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 76 | 86
units on a scale | -0.8 (2.38) | -0.1 (2.64)

10. Secondary Outcome: Difference in Allodynia Rating Between the CRPS-affected Limb and the Normal Limb at Week 12
Description: The investigator rated the degree of allodynia on both the CRPS-affected limb and the normal (or less-affected) limb on an eleven-point scale where 0=no pain and 10=worst pain imaginable. This outcome compares the values for the CRPS affected-limb to the normal limb at week 12.
Time Frame: Week 12
Population: Intent to treat population. Last observation carried forward. Fifteen participants were missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 76 | 87
units on a scale | 3.7 (3.23) | 4.1 (3.41)

11. Secondary Outcome: Change From Baseline in the Brief Pain Inventory (BPI) Total Score at Week 12
Description: Participants completed the Brief Pain Inventory which asks twelve questions that are rated on an eleven-point scale in which 0=most positive outcome and 10=the most negative outcome for a total scale of 0-120. BPI contains questions that concern the level of pain over the last week and the level of pain right now, the extent to which pain interfered with sleep, normal activities, ability to work, relationships, walking etc. Week 12 values are compared to baseline values. Negative change values indicate improvement.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Three participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 85 | 92
units on a scale | -4.8 (13.03) | -3.7 (12.22)

12. Secondary Outcome: Change From Baseline in the Profile of Mood States (POMS) at Week 12
Description: Participants completed the Profile of Mood States questionnaire that asks participants to rate how each of 65 words reflected their mood in the past week on a 5-point scale with 0=not at all and 4=extremely for a total scale of 0-260. Week 12 values are compared to baseline values. Negative change values indicate improvement.
Time Frame: Day 0, week 12
Population: Intent to treat population. Last observation carried forward. Six participants had no post-treatment values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 84 | 90
units on a scale | -9.6 (33.99) | -4.5 (33.91)

13. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 12
Description: The Patient Global Impression of Change asks the question: Overall, how would you rate your CRPS condition since the start of study drug? Answers are represented on a seven-point scale with -3=much worst and +3=much better.
Time Frame: Week 12
Population: Intent to treat. Forty-five participants had no week 12 values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 61 | 74
units on a scale | 0.2 (1.45) | 0.2 (1.41)

14. Secondary Outcome: Participants Who Had a Change to CRPS Pain Medication During the Treatment Period
Description: Participants who had any change in CRPS medication during the double-blind treatment period (up to week 12) are summarized. Changes include additions, discontinuations or dosage change of CRPS medication(s).
Time Frame: Day 1 to week 12
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 87 | 93
participants
  Change to CRPS medication(s) | 11 | 7
  No change to CRPS medication | 76 | 86

15. Secondary Outcome: Change From Baseline in the Maximal Composite Motor Nerve Conduction Velocity at Week 12
Description: An electrophysiological evaluation using standard electrophysiological and electromyography to measure the speed and extent of nerve conduction. Week 12 values are compared to baseline values for maximal motor nerve conduct velocity.
Time Frame: Day 0, week 12
Population: Intent to treat population. Fifty participants did not have week 12 values.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 57 | 73
meters/second | 0.3 (1.56) | 0.1 (2.14)

16. Secondary Outcome: Change From Baseline in the Maximal Composite Sensory Nerve Conduction Velocity at Week 12
Description: An electrophysiological evaluation using standard electrophysiological and electromyography to measure the speed and extent of nerve conduction. Week 12 values are compared to baseline values for maximal sensory nerve conduct velocity.
Time Frame: Day 0, week 12
Population: Intent to treat population. Fifty participants did not have week 12 values.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 56 | 74
meters/second | 1.2 (3.51) | 0.1 (3.41)

17. Secondary Outcome: Participants With Treatment-Emergent Adverse Events in the Double-Blind Period or the Extension Period
Description: Counts of study participants who had adverse events (AEs) while treated in either the Double-blind or Extension Periods. The NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 was used by the investigator to grade the severity of the AEs: Grade 1=Mild AE, Grade 2=Moderate AE, Grade 3=Severe AE, Grade 4=Life-threatening or disabling AE, Grade 5=Death related to AE.
  AEs are also summarized by whether they were serious, related to treatment and whether the AE caused treatment to be altered.
  A serious AE (SAE) was any event that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect or was an important medical event could have jeopardized the patient's safety or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Day 1 up to week 158
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Number analyzed (Participants) | 87 | 93
participants
  Adverse event (AE) | 83 | 85
  Serious adverse event (SAE) | 12 | 16
  AE leading to study drug discontinuation | 29 | 29
  AE leading to dose reduction or interruption | 10 | 8
  Treatment-related AE | 68 | 66
  Treatment-related SAE | 1 | 5
  Grade 2 or higher AE | 63 | 68
  Grade 3 or higher AE | 15 | 18

ADVERSE EVENTS:
Time Frame: Day 1 up to week 158, covering both the double-blind treatment and extension periods.
Description: If multiple SAEs were reported within a given preferred term, only one event was counted per subject.
Arm/Group | Lenalidomide | Placebo to Lenalidomide
Serious Adverse Events (participants affected / at risk) | 12/87 | 16/93
Other Adverse Events (participants affected / at risk) | 77/87 | 72/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=87) | Placebo to Lenalidomide (N=93)
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Thrombosis (Vascular disorders) | 1 | 0
Blood human chorionic gonadotropin positive (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1
Pregnancy test false positive (Investigations) | 1 | 0
Neuropathic pain (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 1
Bradycardia NOS (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Adrenal insufficiency NOS (Endocrine disorders) | 0 | 1
Thyroiditis NOS (Endocrine disorders) | 0 | 1
Cholecystitis NOS (Hepatobiliary disorders) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Pregnancy NOS (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Abortion spontaneous NOS (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemolytic anemia NOS (Blood and lymphatic system disorders) | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 0 | 1
Pain NOS (General disorders) | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 1
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Angioneurotic edema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=87) | Placebo to Lenalidomide (N=93)
Rash NOS (Skin and subcutaneous tissue disorders) | 24 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4
Contusion (Skin and subcutaneous tissue disorders) | 3 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 14 | 15
Diarrhoea NOS (Gastrointestinal disorders) | 11 | 10
Constipation (Gastrointestinal disorders) | 8 | 5
Vomiting NOS (Gastrointestinal disorders) | 5 | 4
Headache (Nervous system disorders) | 9 | 13
Dizziness (Nervous system disorders) | 9 | 6
Fatigue (General disorders) | 9 | 12
Pyrexia (General disorders) | 6 | 4
Fall (General disorders) | 3 | 5
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Urinary tract infection NOS (Infections and infestations) | 3 | 6
Sinusitis NOS (Infections and infestations) | 5 | 3
Alanine aminotransferase increased (Investigations) | 5 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.